CLINICAL TRIAL: NCT00955071
Title: Dose-response Effects of Exercise on Abdominal Obesity and Risk Factors for CVD in Men and Women.
Brief Title: Effects of Exercise on Abdominal Obesity and Risk Factors for Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bob Ross, Ph.D., Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ross 2009
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Obesity; Metabolic Syndrome; Cardiovascular Disease
Keywords: exercise; physical activity; diet; metabolic risk; visceral fat; Insulin Resistance
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Cardiovascular Diseases; Motor Activity; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention)
- Exercise: LVLI (Active Comparator): low volume, low intensity
  Interventions: Other: Exercise: LVLI
- Exercise: HVLI (Active Comparator): high volume, low intensity
  Interventions: Other: Exercise: HVLI
- Exercise: LVHI (Active Comparator): low volume, high intensity
  Interventions: Other: Exercise: LVHI

INTERVENTIONS:
Other: Exercise: LVLI — low volume, low intensity
  Arms: Exercise: LVLI
Other: Exercise: HVLI — high volume, low intensity
  Arms: Exercise: HVLI
Other: Exercise: LVHI — low volume, high intensity
  Arms: Exercise: LVHI

SUMMARY:
The investigators will randomize abdominally obese men and women at increased health risk to one of the following 4 conditions: 1) No-exercise, wait list controls (C), 2) Low volume, low intensity exercise (LVLI), 3) High volume, low intensity exercise (HVLI), 4) Low volume, high intensity exercise (LVHI).

The primary aim of the trial is to determine the effects of varying exercise dose (energy expenditure, kcal) or intensity (relative to VO2max (cardiorespiratory fitness)) on waist circumference and glucose tolerance. The investigators will test the following hypotheses: 1) That the reduction in waist circumference and improvement in glucose tolerance in response to all treatments will be greater than controls. 2) That reduction in waist circumference and improvement in glucose tolerance in HVLI and LVHI will be greater than LVLI. 3) That hypotheses 1 and 2 are true independent of gender.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 40 and 60 years of age. The lower age range for men and women is selected to help ensure recruitment of a sample with metabolic syndrome as prevalence of metabolic syndrome is significantly related to age. The selection of 60 years for the upper age range reflects concerns we have randomizing older adults to the high intensity exercise group wherein exercise at 75-80% of maximum may be difficult to achieve, and likely to be associated with increase orthopaedic injury and thus, poor compliance. We also considered lowering the lower age range from 40 to 35 years, but decided against doing so to increase the cost-effectiveness of recruitment (e.g., ensure a higher yield of those with metabolic syndrome).
* Abdominally obese (waist circumference greater than 88 and 102 cm for women and men respectively) and NCEP-ATPIII defined Metabolic Syndrome. Abdominal obesity for non-Caucasians will be determined using values suggested by the International Diabetes Federation.
* Sedentary lifestyle (planned physical activity for the purpose of health one day per week or less).
* Weight stable (± 2 kg) for 6 months prior to the beginning of the study.
* BMI less than 40 kg/m2 (Because a lifestyle-based intervention alone for obesity reduction is ideal for persons with a BMI less than 40 kg/m2).

Exclusion Criteria:

* Physical impairment which would make the intervention very difficult, or unsafe according to the patient's physician including history of myocardial infarction, stroke, coronary bypass surgery or angioplasty in the last 6 months; peripheral artery disease, unstable angina or ischemia.
* Diabetes.
* Current smokers.
* Alcohol consumption > 21 drinks per week.
* Plans to move from the area.
* Participating in another research study.
* Clinically judged to be unsuitable for participation or adherence as determined by the participants physician.
* Inability or unwillingness to provide informed consent.
* For women, planned pregnancy in the next year.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
waist circumference | 6 months
2-hour glucose | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, PhD, Principal Investigator — Queen's University; Robert Hudson, MD,PhD, Principal Investigator — Queen's University; Miu Lam, PhD, Principal Investigator — Queen's University
Locations (1):
- School of Kinesiology and Health Studies, Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Cowan TE, Brennan AM, Stotz PJ, Clarke J, Lamarche B, Ross R. Separate Effects of Exercise Amount and Intensity on Adipose Tissue and Skeletal Muscle Mass in Adults with Abdominal Obesity. Obesity (Silver Spring). 2018 Nov;26(11):1696-1703. doi: 10.1002/oby.22304. Epub 2018 Sep 27. PMID 30261125
- [Derived] Ross R, Hudson R, Stotz PJ, Lam M. Effects of exercise amount and intensity on abdominal obesity and glucose tolerance in obese adults: a randomized trial. Ann Intern Med. 2015 Mar 3;162(5):325-34. doi: 10.7326/M14-1189. PMID 25732273
- [Derived] Ross R, Hudson R, Day AG, Lam M. Dose-response effects of exercise on abdominal obesity and risk factors for cardiovascular disease in adults: study rationale, design and methods. Contemp Clin Trials. 2013 Jan;34(1):155-60. doi: 10.1016/j.cct.2012.10.010. Epub 2012 Nov 1. PMID 23123790